CLINICAL TRIAL: NCT02309632
Title: Pancreatic Cancer Screening of High-Risk Individuals in Arkansas
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 203640
Record Dates: First submitted 2014-12-03; First posted 2014-12-05 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Pancreatic Neoplasms; Peutz-Jegher's Syndrome; BRCA1 Gene Mutation; BRCA2 Gene Mutation; Ataxia Telangiectasia; Familial Atypical Mole-Malignant Melanoma Syndrome; Colorectal Neoplasms, Hereditary Nonpolyposis; Hereditary Pancreatitis
MeSH Terms: conditions — Pancreatic Neoplasms; Peutz-Jeghers Syndrome; Ataxia Telangiectasia; Melanoma, Cutaneous Malignant; Colorectal Neoplasms, Hereditary Nonpolyposis; Hereditary pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pathway 1 (Active Comparator): Individuals at high risk of pancreatic cancer who will participate in Pancreatic Cancer Screening Pathway 1
  Interventions: Other: Pancreatic Cancer Screening Pathway 1
- Pathway2 (Active Comparator): Individuals at high risk of pancreatic cancer who will participate in Pancreatic Cancer Screening Pathway 2
  Interventions: Other: Pancreatic Cancer Screening Pathway 2

INTERVENTIONS:
Other: Pancreatic Cancer Screening Pathway 1 — Screening with imaging and biomarker testing
  Arms: Pathway 1
Other: Pancreatic Cancer Screening Pathway 2 — Screening with biomarker testing only
  Arms: Pathway2

SUMMARY:
100 subjects who have a family history of pancreatic cancer (PC), or known genetic syndromes associated with increased risk of pancreatic cancer, will be followed for five years. This data will be used to determine the pancreatic cancer and precancerous lesion detection rate in High Risk Individuals (HRIs). Subjects may agree to annual imaging and annual biomarkers or to biomarkers only.

ELIGIBILITY:
Inclusion Criteria:

* Have a family history of PC as listed below or who have one of the following syndromes: Peutz-Jeghers syndrome - STK11; BRCA 1 and 2; PALB2; ATM; FAMMM / P16; HNPCC (Lynch) / MMR genes; Hereditary pancreatitis - PRSS1
* Individuals with three or more affected blood relatives (1st, 2nd or 3rd degree)
* Individuals with two or more affected blood relatives with PC, with at least one affected FDR, should be considered for screening.
* Patients with a history of Peutz-Jeghers syndrome should be screened, regardless of family history of PC.
* Patients with a known p16 (FAMMM syndrome) with one affected 1st or 2nd degree relative will be considered for screening.
* Patients with a known BRCA1 or BRCA2 mutation with one affected 1st or 2nd degree relative should be considered for screening.
* Patients with a known PALB2 mutation with one affected family member should be considered for screening.
* Patients with a known Mismatch-repair gene-mutation carriers (Lynch syndrome) with one affected family member should be considered for screening.

Exclusion Criteria:

* Not candidates for surgery

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11 (Estimated); Primary Completion 2019-07-19 (Actual); Study Completion 2019-07-19 (Actual)

PRIMARY OUTCOMES:
Detection rate of PC and precancerous lesion | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Kent D McKelvey, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States